CLINICAL TRIAL: NCT04493866
Title: Delivering High Quality Documentation on Operative Consent Forms; A UK Major Trauma Centre Quality Improvement Study
Brief Title: Quality Improvement Study on Operative Consent Forms
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 287762
Record Dates: First submitted 2020-07-22; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-05

CONDITIONS: Quality Improvement; Informed Consent

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Messages to departmental employees to improve quality of consent form completion — All interventions directed to members of the plastic surgery department: Intervention 1: Poster illustration common mistakes on consent forms. Intervention 2: Group message explaining Quality Improvement Project to the department. Intervention 3: Email from Consultant lead in support of project. Intervention 4: Further group message illustrating gains and ongoing goals of the project.

SUMMARY:
A Quality Improvement Project was undertaken to improve the completion of operative consent forms within a UK hospital plastic surgery department. Four weekly interventions were made which were accompanied by four further data collection cycles.

DETAILED DESCRIPTION:
Background Royal College of Surgeons guidelines exist on the importance of full, accurate and legible completion of consent forms as a key part of the process of gaining informed consent. In addition to this, consent forms serve as an important medico-legal document to protect clinicians and patients should problems arise. It is therefore in all parties' interests that they are correctly completed.

It was noted that consent forms within the Royal London Hospital Plastic Surgery department were often not correctly completed. A Quality Improvement Project was undertaken to improve the completion of consent forms within the department.

Materials and Methods Common problem areas on consent forms were identified and QI methodology was used to design the study including selection of appropriate outcome, process and balancing measures. Baseline information on completion of: 1) patient details, 2) consultant details, 3) legibility, 4) use of abbreviations in description of operation/complications, and 5) patient signatures was collected. Four weekly interventions were made which were accompanied by four further data collection cycles. A further re-audit took place 4 months following the completion of the project to establish whether improvements had been sustained.

ELIGIBILITY:
Inclusion Criteria:

* Operative Consent form 1 or Consent form 2 completed within the Royal London Hospital Plastic surgery department within one week of the previous intervention.

Exclusion Criteria:

* All other consent forms

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The operative consent form of any adult or paediatric patient consented for an operative procedure within the Royal London Hospital Plastic surgery department within the time frame of the Quality Improvement Project.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Legibility of consent forms | 4 weeks
  Number of operative consent forms that are overall legible (rather than illegible) as assessed by 2 members of the quality improvement team. In cases of differing of opinion on legibility a third member the team to assess.
Full population of patient signature, writing of name and dating of operative consent form | 4 weeks
  Number of operative consent forms with full population of: patient signature + patient writing of name + patient dating of operative consent form
Omission of all abbreviations from written description of operation + risks of operation + benefits of operation on operative consent form | 4 weeks
  Number of operative consent forms with: omission of all abbreviations from written description of operation / risks of operation / benefits of operation fields on operative consent form

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Stodell, FRCS, Study Director — Barts and the Royal London NHS Trust
Locations (1):
- BartsLondonNHS, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
No sharing of participant data will take place.

REFERENCES:
- [Background] Gillon R. Defending the four principles approach as a good basis for good medical practice and therefore for good medical ethics. J Med Ethics. 2015 Jan;41(1):111-6. doi: 10.1136/medethics-2014-102282. PMID 25516950
- See also: 1. Wai Hung Yau et al. Clinical Negligence Costs: taking action to safeguard NHS sustainability. BMJ 2020; 368 doi — https://doi.org/10.1136/bmj.m552
- See also: 2. House of Commons Committee of public accounts. Managing the costs of clinical negligence in hospital trusts. Fifth report of session 2017-2019. (accessed 4th July 2020) — https://publications.parliament.uk/pa/cm201719/cmselect/cmpubacc/397/397.pdf
- See also: 2. House of Commons Committee of public accounts. Managing the costs of clinical negligence in hospital trusts. Fifth report of session 2017-2019. (accessed 4th July 2020) — https://www.rcseng.ac.uk/news-and-events/media-centre/press-releases/surgeons-warn-nhs-failing-to-implement-patient-consent-rules/
- See also: 5. Royal College of Surgeons Guidelines on Good Surgical Practice Sept 2014 section 3.5.1 'Consent'. (accessed 4th July 2020) — https://www.rcseng.ac.uk/standards-and-research/gsp/domain-3/3-5-1-consent/
- See also: 6. Institute for Healthcare Improvement; Quality Improvement Essentials Toolkit. (accessed 4th July 2020) — http://www.ihi.org/resources/Pages/Tools/Quality-Improvement-Essentials-Toolkit.aspx